CLINICAL TRIAL: NCT03111485
Title: Effect of Long-acting Levodopa on Obstructive Sleep Apnea in Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Weston Brain Institute (Other)
Responsible Party: Principal Investigator, Marta Kaminska, Assistant Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP-37-2017-2573
Record Dates: First submitted 2017-03-28; First posted 2017-04-12 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Parkinson's Disease; Obstructive Sleep Apnea
MeSH Terms: conditions — Parkinson Disease; Sleep Apnea, Obstructive | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (drug-placebo) (Experimental): Sinemet CR (Long-acting levodopa: levodopa 200mg/ carbidopa 50mg) followed by a washout period and placebo oral capsule, each taken at bedtime for 2 weeks
  Interventions: Drug: Sinemet CR; Drug: Placebo oral capsule
- B (placebo-drug) (Experimental): Placebo oral capsule followed by a washout period and Sinemet CR (Long-acting levodopa: levodopa 200mg/ carbidopa 50mg), taken at bedtime for 2 weeks
  Interventions: Drug: Sinemet CR; Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Sinemet CR — Capsule 250 mg / 50 mg taken at bedtime
  Other Names: Long acting levodopa
Drug: Placebo oral capsule — Capsule taken at bedtime
  Other Names: Placebo

SUMMARY:
This trial will assess whether long-acting levodopa taken at night improves obstructive sleep apnea (OSA) in patients with Parkinson's disease (PD), as compared with placebo.

DETAILED DESCRIPTION:
Participants with Parkinson's disease and sleep apnea will take long-acting levodopa and placebo at bedtime for 2 weeks each, in a randomized order, with a 2-week washout period in-between. Sleep studies will be done at the end of each period. The primary outcome will be the apnea-hypopnea index change from baseline to on-medication, comparing active medication to placebo. Other outcomes will include other polysomnographic parameters such as oxygenation measures and sleep architecture variables, as well as the Epworth Sleepiness Scale, the Montreal Cognitive Assessment, the Parkinson's disease sleep scale and the Unified Parkinson's Disease Rating Scale. Adverse events will be closely monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic PD consistent with the UK Brain Bank;
2. Presence of OSA on screening PSG, as defined by an AHI ≥ 15/h (moderate to severe OSA);
3. Stable regimen of anti-PD medication for 4 weeks prior to entry into the study, and no planned change during the study

Exclusion Criteria:

1. Other major neurological disorder;
2. Already taking long-acting levodopa (at any time of day);
3. Taking short-acting levodopa at bedtime or during the night;
4. Any contraindication to long-acting levodopa (see below);
5. Severe levodopa induced dyskinesias;
6. Already on or requiring treatment for restless legs syndrome ;
7. Body mass index >35 kg/m2;
8. Intercurrent upper respiratory tract infection;
9. Other known cause of OSA (e.g. craniofacial malformation);
10. Active treatment of OSA (CPAP, dental appliance or other), unless willing to stop treatment 2 weeks prior to start and during the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Apnea-hypopnea index (AHI) | 2 weeks

SECONDARY OUTCOMES:
Proportion of patients having adverse events leading to discontinuation of drug (Feasibility and tolerability) | 2 weeks
  Proportion of patients having adverse events leading to discontinuation of drug
Oxygenation from polysomnography | 2 weeks
  oxygen desaturation index
Oxygenation from polysomnography | 2 weeks
  mean oxygen saturation
Oxygenation from polysomnography | 2 weeks
  time with saturation below 90%
Objective sleep quality from polysomnography | 2 weeks
  Sleep efficiency
Objective sleep quality from polysomnography | 2 weeks
  total sleep time
Objective sleep quality from polysomnography | 2 weeks
  wake after sleep onset
Objective sleep quality from polysomnography | 2 weeks
  sleep stages distribution
Objective sleep quality from polysomnography | 2 weeks
  arousal index
Subjective sleep quality | 2 weeks
  Parkinson's Disease Sleep Scale-R
Daytime sleepiness | 2 weeks
  Epworth Sleepiness Scale
Non-motor symptoms | 2 weeks
  MDS-UPDRS part I
Cognitive function | 2 weeks
  Montreal Cognitive Assessment (MoCA)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Kaminska, MD, MSc, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No